CLINICAL TRIAL: NCT07333196
Title: Tongji NADs Cohort: A Real-world Observation of Neurological Autoimmune Disorders
Brief Title: Tongji NADs Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Shenzhen Genocury Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Daishi Tian, Professor, Tongji Hospital
Other Study IDs: NADsinTJ
Record Dates: First submitted 2025-12-09; First posted 2026-01-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; NMO Spectrum Disorder; Autoimmune Encephalitis; Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease; Autoimmune Nodopathy; Acute Inflammatory Demyelinating Polyradiculoneuropathy; Chronic Inflammatory Demyelinating Polyradiculoneuropathy; Myasthenia Gravis; Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Autoimmune Diseases of the Nervous System; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Guillain-Barre Syndrome; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Myasthenia Gravis; Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No active interventions — The therapies are based on needs of the participants

SUMMARY:
Neurological Autoimmune Diseases (NADs) are disorders caused by abnormal immune system attacks on neural tissues, affecting multiple systems including the central nervous system, peripheral nervous system, and neuromuscular junctions. This study examines clinically significant NADs such as multiple sclerosis (MS), neuromyelitis optica spectrum disorders (NMOSD), myelin oligodendrocyte glycoprotein G antibody-related diseases (MOGAD), autoimmune encephalitis (AE), immune-mediated peripheral neuropathy (PN), myasthenia gravis (MG), and idiopathic inflammatory myopathy (IIM). While sharing the core pathogenesis of autoimmune response, these diseases exhibit significant heterogeneity in epidemiological patterns, clinical manifestations, therapeutic approaches, and disease progression. This heterogeneity stems from multiple factors: (1) Differences in immune targets: MS primarily involves T-cell-mediated myelin attack, NMOSD is mainly driven by astrocyte damage caused by anti-AQP4 antibodies, MOGAD results from myelin surface loss mediated by antibodies against myelin oligodendrocyte glycoprotein immunoglobulin G, while AE involves synaptic dysfunction due to antibodies against neuronal surface proteins (e.g., anti-NMDA-R antibodies); (2) Genetic-environmental interactions: MS is more prevalent in European and American populations, whereas NMOSD is more aggressive in Asian populations; (3) Variability in treatment response: Some diseases respond well to immunomodulatory therapy, but most still face challenges such as high relapse rates, progressive disability accumulation, and irreversible neurological damage.

While randomized controlled trials (RCTs) provide high-quality core evidence for drug registration, their strict inclusion/exclusion criteria, relatively homogeneous patient populations, and short-term observation designs often fail to fully capture the complex disease progression and treatment response patterns in real-world clinical settings. Additionally, long-term RCTs are frequently constrained by economic factors and sustainability challenges. Therefore, conducting comprehensive real-world observational studies (RWS) on NADs-integrating multi-disease cohorts, long-term follow-up data, and diverse clinical practices-holds significant scientific and clinical value for optimizing treatment strategies and improving long-term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following eligibility criteria at the time of screening to participate in this study.

1.1. The subject is able to understand the purpose and risks of the study, provide informed consent and authorize the use of confidential health information in accordance with national and local privacy regulations.

1.2. Open to both men and women, aged 18-80 years (inclusive) at the time of informed consent.

1.3. Must be diagnosed with one of the following conditions:

1.3.1. This study adhered to the 2017 McDonald criteria for diagnosing multiple sclerosis:

1. ≥2 clinical episodes with ≥2 objective clinical evidences of lesions.
2. ≥2 clinical episodes with one clear historical evidence of the lesion involving specific anatomical site.
3. ≥2 clinical episodes with objective clinical evidence of one lesion, and spatial multiplicity confirmed by clinical episodes in different CNS sites or MRI findings.
4. A single episode with ≥2 objective clinical evidences, confirmed by additional clinical episodes or MRI showing temporal multiple lesions or OCB positivity.
5. A single episode with one objective clinical manifestation, confirmed by clinical seizures or MRI scans across multiple CNS regions to demonstrate spatial multiplicity, and further supported by additional clinical episodes or MRI findings to confirm temporal multiplicity or OCB positivity.
6. Indication for the progressive multifocal sclerosis (PPMS) phase: Disease progression at 1 year (confirmed retrospectively or prospectively), with two of the following three criteria: [1] Spatially multifocal evidence of brain lesions: ≥1 T2-weighted lesion in characteristic MS regions (periventricular, corticoprotuberant, or subarachnoid) [2] Spatially multifocal evidence of spinal lesions: ≥2 T2-weighted lesions in the spinal cord [3] OCB positivity.

1.3.2. This study adhered to the 2015 IPND diagnostic criteria for adult neuromyelitis optica spectrum disorders:

1. NMOSD diagnosis with AQP4-IgG positivity: meeting ≥1 core clinical feature, confirmed by reliable AQP4-IgG detection (CBA method recommended), and excluding other diagnoses.
2. Diagnostic criteria for NMOSD with AQP4-lgG negative or undetermined status: In at least one clinical episode, the presence of ≥2 core clinical features meeting all of the following criteria: ①≥1 core clinical feature is ON, acute LETM, or bulbar syndrome; ②≥2 distinct core clinical features; ③MRI supplementary criteria are satisfied. AQP4-lgG should be reliably detected as negative or undetected, and other diagnoses must be excluded.

Note: Core clinical features include six cardinal signs: optic neuritis (ON), acute myelitis (LETM), and the final area syndrome (unexplained paroxysmal hiccups, nausea, and vomiting); other brainstem syndromes; symptomatic narcolepsy/hypothalamic syndrome with characteristic hypothalamic MRI lesions; and brain syndrome with characteristic cerebral MRI lesions.

MRI diagnostic criteria: Acute optic neuritis (ON) requires MRI demonstrating one of the following: ① Normal brain MRI or non-specific white matter lesions; ② Long T-weighted signal or T-weighted enhancement exceeding 1/2 of optic nerve length, or optic chiasm involvement; ③ Acute myelitis (LETM) requires three or more consecutive vertebral segments with spinal cord lesions, or spinal cord atrophy exceeding three consecutive vertebral segments in patients with myelitis history; ④ Final region syndrome: lesions in the dorsal medulla or final region. Acute brainstem syndrome: periventricular lesions in the brainstem.

1.3.3. This study adhered to the MOGAD diagnostic criteria established by the International Parkinson's Disease and Movement Disorders (IPMD) in 2023:

1. A diagnosis of MOGAD can be confirmed when: (a) fixed or live-cell CBA detects strong positivity of MOG-IgG in serum with ≥1 core clinical manifestation, and (b) other diagnoses (e.g., MS, NMOSD) are excluded;
2. If the CBA shows weak positivity of MOG-IgG in serum, or MOG-IgG positivity without titer, or negative serum MOG-IgG with strong positivity in cerebrospinal fluid (CSF), the diagnosis requires: 1) ≥1 core clinical manifestation, 2) ≥1 supporting clinical or imaging feature, 3) negative serum AQP4-IgG, and 4) exclusion of other diagnoses (e.g., MS, NMOSD).

Note: The core clinical features include six main signs: optic neuritis, myelitis, acute disseminated encephalomyelitis, monofocal or multifocal cerebral dysfunction, brainstem or cerebellar functional deficits, and cerebral cortex inflammation with epilepsy.

Typical MRI imaging features: ① Optic Neuropathy (ON): Bilateral optic nerve involvement with long-segment optic nerve damage (>50% optic nerve length), optic nerve sheath enhancement, and papilledema. ② Myelitis: Long-segment transverse myelitis with central spinal cord damage or "H" sign, and conus medullaris damage. ③ Cerebral, brainstem, or cerebral cortex symptoms: Multifocal ill-defined T2 hyperintense lesions in supratentorial and infratentorial white matter, deep gray matter involvement, ill-defined T2 hyperintense lesions in pons, cerebellar midfoot, or medulla oblongata, and cortical lesions with or without focal enhancement and local dural enhancement.

The strong positive result of serum and cerebrospinal fluid MOG-IgG was defined as the value of the live CBA was more than 2 times the detection limit or the fixed CBA titer was ≥1:100. The weak positive result was defined as the value of the live CBA was in the lower range or the fixed CBA titer was ≥1:10 but less than 1:100.

1.3.4. This study followed the expert consensus on the diagnosis and treatment of autoimmune encephalitis in China (2022 edition)

1. Possible AE: meeting the following three diagnostic criteria A, B, and D; confirmed AE: meeting the four diagnostic criteria A, B, C, and D.
2. Diagnostic criteria:

A. Clinical presentation: Acute or subacute onset (<3 months) with ≥1 of the following neurological or psychiatric symptoms or clinical syndromes: limbic system symptoms, encephalitis syndrome, lymphocytic inflammation in cerebrospinal fluid cytology, and positive specific oligoclonal bands.

B. Neuroimaging or electrophysiological abnormalities: T2 or FLAIR abnormal signals in the limbic system (unilateral or bilateral), or T2/FLAIR abnormalities in other regions (excluding nonspecific white matter changes and stroke); or PET findings of high metabolism in the limbic system, or multiple high metabolic areas in the cortex and/or basal ganglia; or EEG abnormalities such as focal epilepsy or epileptiform discharges (in the temporal lobe or outside it), or diffuse or multifocal slow-wave rhythms.

C. Diagnostic test: Positive for anti-neuronal antibodies. D. Reasonably rule out other possible causes.

1.3.5. This study adhered to the diagnostic criteria for AIDP, CIDP, and autoimmune Ranvier node disease:

1. AIDP: Essential features include: ① Progressive weakness in the upper and/or lower limbs, ranging from mild bilateral lower limb weakness to complete paralysis of all limbs (including trunk, medullary muscles, and facial muscles) and oculomotor muscle paralysis; ② Weakened or absent deep tendon reflexes in the affected limbs; ③ Symptom progression ≤4 weeks. Supporting features include: ① Symptom progression from days to 4 weeks; ② Relatively symmetrical bilateral symptoms; ③ Trunk or limb pain; ④ Cranial nerve symptoms or signs; ⑤ Autonomic dysfunction; ⑥ Respiratory insufficiency; ⑦ Mild or absent sensory dysfunction; ⑧ History of prodromal systemic infection in approximately 70% of cases; ⑨ No fever at symptom onset; ⑩ Elevated cerebrospinal fluid protein with normal or mildly elevated white blood cell count (<5 mm³); ⑪ Electrophysiological examination showing abnormalities consistent with Guillain-Barré syndrome (GBS); ⑫ Recovery begins 2-4 weeks after symptom stabilization.
2. CIDP: CIDP develops in 2%-5% of patients initially diagnosed with AIDP, with the following clinical features: ① Progressive or recurrent disease progression lasting over 8 weeks; ② Only approximately 30% of patients experience prodromal events; ③ Additional supporting features include: ≥3 acute relapses or exacerbations occurring ≥8 weeks after symptom onset, milder symptoms, preserved independent walking ability throughout the disease course, and absence of cranial nerve involvement or frequent respiratory system involvement.
3. Autoimmune Ranvier node disease:

   * Clinical manifestations: a. Acute, subacute or chronic course, with persistent progression after 8 weeks of onset; b. Clinical features consistent with polyneuropathy; c. May be accompanied by significant ataxia, tremor or neuropathic pain; d. May be associated with nephrotic syndrome.
   * Electrophysiological findings: a. Motor nerve conduction tests reveal prolonged distal motor latency, slowed conduction velocity, abnormal waveform dispersion, and conduction block, with decreased F-wave conduction velocity, consistent with myelination abnormalities; b. Both motor and sensory nerve conduction show markedly reduced amplitude. Electromyography (EMG) at needle electrodes demonstrates abnormal spontaneous potentials and decreased recruitment, indicating early axonal damage.
   * Antibody detection: serum anti-Langfei junction antibody was positive, especially serum anti-NF155, anti-CNTN1, anti-Casp1 and anti-NF140/186 antibody.
   * Cerebrospinal fluid (CSF) analysis: Protein-cell dissociation is observed, with CSF protein levels typically showing significant elevation.

1.3.6. This study adheres to the diagnostic criteria of the 2024 China Expert Consensus on the Diagnosis and Treatment of Refractory Systemic Myasthenia Gravis

1. Basic conditions

   ① Meet the diagnostic criteria in the China Guidelines for the Diagnosis and Treatment of Myasthenia Gravis (2025 edition).

   ② The patient's Myasthenia Gravis Activities of Daily Living (MG-ADL) score was ≥6, and the ocular muscle score was less than 50% of the total score.
2. Diagnostic criteria:

   * After adequate duration of treatment with at least two conventional immunotherapeutic agents (including both corticosteroids and non-corticosteroid immunosuppressants), the post-intervention status (PIS) remains unchanged or worsens.
   * After adequate doses and duration of at least two conventional immunotherapeutic drugs, the PIS showed improvement, but the MG-ADL score remained ≥6 points for at least six months.
   * After adequate duration of treatment with at least two conventional immunotherapeutic agents, the PIS was remitted or improved, but during the regular tapering of immunotherapy, disease symptoms worsened ≥2 times per year (MG-ADL score ≥6).
   * Patients who, after a crisis, received multiple immunotherapies including intravenous immunoglobulin (IVIG), plasma exchange, and high-dose intravenous methylprednisolone (IVMP), along with active infection control, still remained unable to wean off mechanical ventilation for more than 14 days due to MG-induced respiratory muscle weakness.

Diagnostic criteria: meeting all the above basic conditions plus 1 of the 4 diagnostic conditions.

1.3.7. This study adheres to the 2017 diagnostic criteria for idiopathic inflammatory myopathy (IIM) established by the European League Against Rheumatism (EULAR) and the American College of Rheumatology (ACR), following the EULAR/ACR classification system. Patients with a probability score ≥55% in the table below are considered suspected IIM cases. Suspected IIM patients can be diagnosed with dermatomyositis in adults if they meet the following criteria: ① Age ≥18 years at first onset of IIM-related symptoms; ② Presence of Heliotrope sign, Gottron papules, or Gottron sign; ③ Objective proximal symmetrical arm weakness (confirmed by manual muscle strength testing or other strength assessment methods), typically progressive, or objective proximal symmetrical leg weakness, typically progressive, or more pronounced neck flexor weakness than neck extensor weakness, or more pronounced proximal leg weakness than distal leg weakness. If patients meet criteria ① and ② but not ③, they may be diagnosed with non-myopathic dermatomyositis. Compared to previous standards, this criterion demonstrates higher sensitivity and specificity. In this standard, patients with typical clinical manifestations (such as characteristic rashes) do not require further tests (e.g., muscle biopsy), while some patients without typical rashes may be missed.

Exclusion Criteria:

* This is an observational study with no specific exclusion criteria.
* The investigators identified other unexplained factors that may have disqualified participants from enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to enroll NADs patients meeting inclusion criteria at our center from March 1, 2022 to March 1, 2032. The planned retrospective and prospective cohort will include: 300 multiple sclerosis (MS) cases, 300 AQP4 antibody-positive neuromyelitis optica spectrum disorders (NMDs), 200 MOG antibody-associated diseases, 150 autoimmune encephalitis (AE) cases, 80 immune-mediated peripheral neuropathy (IMPN) cases, 400 myasthenia gravis (MG) cases, and 120 idiopathic inflammatory myopathy (IIM) cases.
Sampling Method: Non-Probability Sample
Enrollment: 1550 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2036-03-01 (Estimated); Study Completion 2037-03-01 (Estimated)

PRIMARY OUTCOMES:
EDSS Score | 10 years from the date of enrollment
  EDSS Score is the most commonly used in evaluating the neurological functions of patients with central nervous system demyelination. The range is 0-10.0.
modified Rankin Score | 10 years from the date of enrollment
  Modified Rankin score is the most commonly used in evaluating the daily life ability of patients with neurological disorders. The range is 0-6.
MMT-8 Score | 10 years from the date of enrollment
  MMT-8 Score is mostly used in evaluating muscle strength of patients with myopathy. The range is 0-150.
QMG Score | 10 years from the date of enrollment
  An authoritative quantitative scale to assess the disease severity of patients with myasthenia gravis. The range is 0-39.
Annual recurrence rate | 10 years from the date of enrollment
Adverse event | 10 years from the date of enrollment
  All participants with treatment-related adverse events as will be assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Quantification of pathogenic antibodies | 10 years from the date of enrollment
  Typical pathogenic antibodies include anti-AQP4-IgG, anti-MOG-IgG, anti-GFAP-IgG, anti-NMDAR-IgG, anti-LGI1-IgG, anti-AMPA-IgG, anti-AchR-IgG, anti-MUSK-IgG, etc, which are tested by ELISA in mmol/l.
Quantification of cytokines | 10 years from the date of enrollment
  Common cytokines include IL2, IL2R, IL6, IL8, IL10, TNFα, etc.
Quantitative and qualitative analysis of immunocyte subtypes | 10 years from the date of enrollment
  Common subtypes include CD3+CD19-,CD3-CD19+,CD3+CD4+,CD3+CD8+,CD3-CD16+CD56+,CD3+CD56+, etc. They are showed in cells/ul.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China